CLINICAL TRIAL: NCT07295691
Title: Autologous Serum Eye Drops in Dry Eye Syndrome: Clinical Efficacy and Safety Evaluation
Brief Title: Autologous Serum Eye Drops in Dry Eye Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The General Authority for Teaching Hospitals and Institutes (Network)
Responsible Party: Principal Investigator, Hossam Abdelfattah Husein Hassan, Fellow of Ophthalmology, Sohag Teaching Hospital, Egypt., The General Authority for Teaching Hospitals and Institutes
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSO00010
Record Dates: First submitted 2025-12-06; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Autologous Serum Eye Drops; Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Participants will receive eye drops prepared from their blood serum following a standardized protocol. Specifically, 40 mL of venous blood was collected from each participant at the start of the study and centrifuged at 3000 rpm for 15 min.
  Interventions: Other: Autologous Serum Eye Drop

INTERVENTIONS:
Other: Autologous Serum Eye Drop — Participants will receive eye drops prepared from their blood serum following a standardized protocol. Specifically, 40 mL of venous blood was collected from each participant at the start of the study and centrifuged at 3000 rpm for 15 min.

SUMMARY:
This study aims to evaluate the clinical efficacy and safety of autologous serum eye drops (ASEDs) in patients with moderate-to-severe dry eye syndrome who are refractory to conventional artificial tear therapy.

DETAILED DESCRIPTION:
Dry Eye Syndrome (DES) is a highly prevalent ocular condition that significantly affects quality of life, with global prevalence estimated at 5%-50%, depending on population and diagnostic criteria.

Autologous Serum Eye Drops (ASEDs) have emerged as a promising therapy due to their composition, which is rich in vitamin A, epidermal growth factor, fibronectin, and transforming growth factor-β. These components mimic natural tears and promote epithelial healing, reduce inflammation, and enhance tear film stability.

ELIGIBILITY:
Inclusion Criteria:

* Children aged less than 18 years.
* Both sexes.
* Diagnosed with moderate to severe dry eye syndrome (DES) refractory to artificial tears.

Exclusion Criteria:

* Active ocular infection.
* Recent ocular surgery.
* Systemic immunosuppressive therapy.
* History of allergy to blood-derived products.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 12 weeks post-procedure
  Visual acuity will be measured.

SECONDARY OUTCOMES:
Improvement in Ocular Surface Disease Index (OSDI) | 12 weeks post-procedure
  The ocular surface disease index (OSDI) is a comprehensive 12-item questionnaire used to assess the frequency and severity of eye symptoms, the influence of environmental triggers, and the impact of DES on vision-related functionality. The OSDI scores range from 0 to 100, with higher scores indicating greater ocular discomfort and impairment.
Incidence of adverse events | 12 weeks post-procedure
  Incidence of adverse events will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- The General Authority for Teaching Hospitals and Institutes, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.